CLINICAL TRIAL: NCT02056704
Title: A Prospective Randomized Feasibility Trial Comparing Angiography and Angiography With IVUS for Treatment of Hemodialysis Access Failures
Brief Title: Trial Comparing Angiography and Angiography With IVUS for Treatment of Hemodialysis Access Failures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 012-088
Record Dates: First submitted 2014-01-29; First posted 2014-02-06 (Estimated); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Dialysis Access Malfunction
Keywords: Dialysis Fistula; Dialysis Graft; Stenosis; Intravascular Ultrasound; Angiography
MeSH Terms: conditions — Constriction, Pathologic | interventions — Angiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Angiography (No Intervention): Evaluation by angiography only.
- Angiography with IVUS (Experimental): Evaluation with angiography and intravascular ultrasound.
  Interventions: Device: Angiography with IVUS

INTERVENTIONS:
Device: Angiography with IVUS — The use of IVUS to evaluate dialysis access failure.
  Other Names: Volcano IVUS catheter
  Arms: Angiography with IVUS

SUMMARY:
The reason the investigators are doing this study is to compare the results of angiography versus angiography with intravascular ultrasound in dialysis grafts/fistulas that are blocked.

DETAILED DESCRIPTION:
Patients with kidney failure have a fistula or graft for long-term dialysis in order for the dialysis machine to draw blood, filter it, and give it back to the patient. Over time, the fistula or graft may not work well enough to use for dialysis, most commonly because the veins may develop "scar tissue" within and around them that narrows the vein resulting in poor flow or complete blockage.

These blockages are commonly opened with wires, balloons (a procedure called angioplasty), and stents. These blockages are seen with angiography, a special type of x-ray used with a dye that shows the inside of the blood vessels. Intravascular ultrasound (IVUS) is a type of imaging that uses sound waves to produce an image of the inside of blood vessels and to see their condition. Currently, it is not known if angiography alone or angiography with IVUS has better results. The reason we are doing this study is to compare the results of angiography versus angiography with IVUS.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* Male or female (non-pregnant females)
* Patients with hemodialysis access failure (arteriovenous fistulae or arteriovenous grafts)
* Patients must undergo elective angiographies (fistulograms) based on surveillance duplex ultrasound findings (stenosis)
* Patients with outflow stenoses between 1 cm distal to an arterial anastamosis and clavicle in AV fistulae or between venous anastamosis and clavicle in AV grafts found on surveillance duplex ultrasound

Exclusion Criteria:

* Patients with other etiologies (inflow lesions, intragraft lesions, hypercoagulable states, lesions not readily amenable to stenting), advanced failures (thrombosis, central venous occlusion), and non-routine access conformations (chest wall/groin grafts, balloon assisted maturation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-02-18 (Actual); Primary Completion 2017-10-20 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Change in characteristics of lesion within the vessel | every 3 months - up to 2 years
  This will include vessel diameters proximal and distal to lesions, percent stenosis, and lesion lengths.

CONTACTS AND LOCATIONS:
Overall Officials: William Shutze, MD, Principal Investigator — Baylor Health Care System
Locations (4):
- United States (4):
  - Baylor Jack and Jane Hamilton Heart and Vascular Hospital, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
  - Baylor Regional Medical Center at Plano, Plano, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas